CLINICAL TRIAL: NCT04666779
Title: Access to Chiropractic Care During the COVID-19 Pandemic: a Prospective Comparative Cohort Trial
Brief Title: Access to Chiropractic Care During the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Real Centro Universitario Maria Cristina (Other)
Collaborators: University of Birmingham (Other); Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other); Université du Québec à Trois-Rivières (Other)
Responsible Party: Sponsor
Other Study IDs: CohortChiroCOVID19
Record Dates: First submitted 2020-12-11; First posted 2020-12-14 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Access to Chiropractic Care Services

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No access: Group not accessing chiropractic care
- Access to care: Group with access to care in a 6 months period. Differences in the degree of access, measured in ranges of numbers of visits, will be used as independent variable within this group.
  Interventions: Other: Chiropractic care

INTERVENTIONS:
Other: Chiropractic care — Care provided by chiropractors, based on manual therapy, exercise prescription and patient advice/education/reassurance
  Groups: Access to care

SUMMARY:
This is a prospective comparative cohort trial taking place during the first year of the Coronavirus-19 (COVID-19) pandemic in Spain. Chiropractic patients throughout Spain were invited to participate independently of the care received, including patients who had stopped visiting their chiropractors since the pandemic hit. The main exposure variable is the access to chiropractic care services, and the degree of this exposure during the months following initial lockdown phase in Spain. Participants will fill an online questionnaire with self-reported outcome-measures.

ELIGIBILITY:
Inclusion Criteria:

* chiropractic patients with pain, active when lockdown was declared, over the age of 16

Exclusion Criteria:

* new patients in the clinic after the pandemic hit

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chiropractic patients when the pandemic hit in Spain (March 2020), who consulted a chiropractor for pain as one of the chief complaints (not necessarily the main or the only one)
Sampling Method: Non-Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 6 months
  Numerical Rating Scale (0-10, 0=no pain, 10=maximum pain)
Pain duration | 6 months
  Duration of pain symptoms, PREVIOUS to the study, measured in months (up to 3 months, more than 3 months)
Pain frequency | 6 months
  Ranges: Constant, every day, every week, occasionally
Pain perceived improvement | 6 months
  Categories: New pain, worsened, no change, improv, gone
Pain interference | 6 months
  From the Brief Pain Inventory (7 items, 0-10: 0= minimal score, 70=maximal score)
Pain Catastrophizing Scale | 6 months
  Validated questionnaire (short version 4 items, 1-4: 4= minimal score, 16=maximal score)
Tampa Scale Kinesiophobia | 6 months
  Validated questionnaire (short version 11 items, 0-3: 0=minimal score, 33=maximal score)

SECONDARY OUTCOMES:
General Anxiety Disorder scale | 6 months
  Validated questionnaire (7 items , 1-3: 1= minimal score, 21=maximal score)
Fear of Illness and Virus Evaluation | 6 months
  Questionnaire (12 items, 1-4: 1=minimal score, 48=maximal score)

CONTACTS AND LOCATIONS:
Overall Officials: Arantxa Ortega de Mues, PhD, Principal Investigator — Real Centro Universitario María Cristina
Locations (1):
- Real Centro Universitario María Cristina, El Escorial, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
All collected IPD will be shared, the format is yet to be decided.